CLINICAL TRIAL: NCT01994616
Title: Intralesional Cryotherapy for Treatment of Keloid Scars: a Prospective Evaluation
Brief Title: Prospective Evaluation of the Use of Intralesional Cryotherapy for Treatment of Keloid and Hypertrophic Scars
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Red Cross Hospital Beverwijk (Other)
Responsible Party: Principal Investigator, Michiel van Leeuwen, Medical Doctor, Amsterdam UMC, location VUmc
Other Study IDs: 12/292
Record Dates: First submitted 2013-11-19; First posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Keloid; Cicatrix, Hypertrophic
Keywords: Keloid, hypertrophic scar
MeSH Terms: conditions — Keloid; Cicatrix, Hypertrophic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- keloid or hypertrophic scars: All patient including all skin types with keloid or hypertrophic disease receiving Intralesional Cryotherapy
  Interventions: Procedure: Intralesional cryotherapy

INTERVENTIONS:
Procedure: Intralesional cryotherapy — Intralesional (IL) cryotherapy is a treatment for keloids and hypertrophic scars, in which the scar is frozen from inside with the use of a cryoneedle
  Other Names: Cryoneedle (CryoShape, Etgar Group International Ltd, Kfar Saba, Israel)

SUMMARY:
This prospective evaluation studies the effectiveness of IL cryotherapy in treating keloids and hypertrophic scars in a large population of mixed Fitzpatrick skin types.

DETAILED DESCRIPTION:
Intralesional (IL) cryotherapy is a novel treatment for keloids and hypertrophic scars, in which the scar is frozen from inside. Published results are promising, however only Caucasian patient populations have been studied. This prospective evaluation studies the effectiveness of IL cryotherapy in treating keloids and hypertrophic scars in a large population of mixed Fitzpatrick skin types. All patients with keloid or hypertrophic scars meeting inclusion criteria were treated with a liquid nitrogen based device called Cryoshape Scar quality and possible recurrence are assessed pre- and postsurgery (3, 6 and 12 months) with objective devices determine scar color, scar elasticity, scar volume and patient's skin type. In addition, scars are evaluated using the Patient and Observer Scar Assessment Scale.

ELIGIBILITY:
Inclusion Criteria:

* Keloids, defined as excessive scar tissue raised above skin level and proliferating beyond the confines of the original lesion
* Hypertrophic scars1 older than 12 months and insensitive to other treatments. Keloids were distinguished from hypertrophic scars based on the clinical judgment of experienced plastic surgeons and on the age of the scar (>1yr)
* A period between previous treatment and IL cryotherapy covered a minimum of 12 weeks
* Patients with all Fitzpatrick17 skin types
* Patients older than 10 years of age

Exclusion Criteria:

* pregnancy
* diabetes mellitus

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A mixed patient population with all Fitzpatrick skin types
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Recurrence | 0-12 months
  Judgment of recurrence, defined as a growing, pruritic, nodular scar

SECONDARY OUTCOMES:
Scar elasticity | 0-12months
  Scar elasticity, measured in two parameters: extension and elasticity

OTHER OUTCOMES:
Scar volume | 0-12months
  Determined by creating a mold of the scar with dental putty
Redness (erythema) and pigmentation (melanin), | 0-12months
  Redness (erythema) and pigmentation (melanin), which were measured using the DermaSpectrometer
Subjective scar evaluation | 0-12months
  performed by two experienced medical doctors and the patient using the Patient and Observer Scar Assessment Scale (POSAS). Each item of the POSAS was scored using a 10-step score, in which 10 reflected 'worst scar imaginable' and 1 indicated 'normal skin'

CONTACTS AND LOCATIONS:
Overall Officials: Michiel CE van Leeuwen, MD, Principal Investigator — VUmc; Frank B Niessen, PhD, MD, Study Director — Vumc
Locations (1):
- VUmc, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Har-Shai Y, Amar M, Sabo E. Intralesional cryotherapy for enhancing the involution of hypertrophic scars and keloids. Plast Reconstr Surg. 2003 May;111(6):1841-52. doi: 10.1097/01.PRS.0000056868.42679.05. PMID 12711943
- [Derived] van Leeuwen MCE, van der Wal MBA, Bulstra AJ, Galindo-Garre F, Molier J, van Zuijlen PPM, van Leeuwen PAM, Niessen FB. Intralesional cryotherapy for treatment of keloid scars: a prospective study. Plast Reconstr Surg. 2015 Feb;135(2):580-589. doi: 10.1097/PRS.0000000000000911. PMID 25626801
- See also: homepage VU medical center, hospital Amsterdam, the Netherlands — http://www.vumc.nl